CLINICAL TRIAL: NCT05825326
Title: Epidemiological and Clinical-pathological Factors of Philadelphia-negative Myeloproliferative Neoplasms in Ecuador
Status: Completed | Type: Observational
Sponsor: Sociedad de Lucha Contra el Cáncer del Ecuador (Other)
Responsible Party: Sponsor
Other Study IDs: CISOLGYE20230022
Record Dates: First submitted 2023-03-27; First posted 2023-04-24 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Myeloproliferative Neoplasm; Myeloproliferative Syndrome; Myeloproliferative Neoplasm, Unclassifiable; Myeloproliferative Disorders; Myeloproliferative Disease, Not Classified
Keywords: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with Philadelphia-negative Myeloproliferative Neoplasms

SUMMARY:
The goal of this observational study is to evaluate the epidemiological and clinical-pathological features of Philadelphia-negative myeloproliferative neoplasms through data from medical records

DETAILED DESCRIPTION:
The investigators are proposing a study that provides descriptive understanding of patients with Philadelphia-negative myeloproliferative neoplasms in Ecuador. The primary objective of this pilot study is to lay the foundations for the development of a multicenter registry of Philadelphia-negative myeloproliferative neoplasms, which will provide high-quality real data and serve as a basis for the application to future projects and elaboration of public policies in the medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients with confirmed diagnosis of Philadelphia-negative Myeloproliferative Neoplasms

Exclusion Criteria:

* Patients with translocation t(9;22)(q34:q11.2) with subsequent formation of the BCR-ABL1 fusion gene determined by cytogenetics or fluorescence in situ hybridization (FISH)
* Absence of the histopathological report in the clinical history and the corresponding plaque, except in the case of Polycythemia Vera that does not require them for diagnosis, according to the 2022 WHO classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Philadelphia-negative Myeloproliferative Neoplasms according to the 2022 World Health Organization (WHO) classification
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with Philadelphia-negative Myeloproliferative Neoplasms in Ecuador | 96 months
  Participants were followed-up for 8 years. This is the number of participants who have had Philadelphia-negative Myeloproliferative Neoplasms in Ecuador during the time of observation.

SECONDARY OUTCOMES:
Prevalence of Philadelphia-negative myeloproliferative patients | 96 months
  Calculation of the prevalence of participants who have had Philadelphia-negative Myeloproliferative Neoplasms in Ecuador during the time of observation.
Mortality risk as measured by the Dynamic International Prognostic Scoring System | 96 months
  The Dynamic International Prognostic Scoring System (DIPSS) was proposed and validated by Passamonti and is used as a prognostic model to predict survival in participants with Primary Myeloid Fibrosis a Philadelphia-negative myeloproliferative neoplasm.
  Possible scores range from 0 to 6, with higher scores indicating higher mortality risk.
Overall survival | 96 months
  Percent of participants with Primary Myeloid Fibrosis who were alive at 96 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fuad Huamán Garaicoa, MD, Principal Investigator — Sociedad de Lucha Contra el Cáncer del Ecuador
Locations (1):
- Sociedad de Lucha Contra el Cáncer, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nangalia J, Green AR. Myeloproliferative neoplasms: from origins to outcomes. Blood. 2017 Dec 7;130(23):2475-2483. doi: 10.1182/blood-2017-06-782037. PMID 29212804
- [Background] Heppner J, Nguyen LT, Guo M, Naugler C, Rashid-Kolvear F. Incidence of myeloproliferative neoplasms in Calgary, Alberta, Canada. BMC Res Notes. 2019 May 24;12(1):286. doi: 10.1186/s13104-019-4321-1. PMID 31126326
- [Background] Hultcrantz M, Kristinsson SY, Andersson TM, Landgren O, Eloranta S, Derolf AR, Dickman PW, Bjorkholm M. Patterns of survival among patients with myeloproliferative neoplasms diagnosed in Sweden from 1973 to 2008: a population-based study. J Clin Oncol. 2012 Aug 20;30(24):2995-3001. doi: 10.1200/JCO.2012.42.1925. Epub 2012 Jul 16. PMID 22802311
- [Background] Roaldsnes C, Holst R, Frederiksen H, Ghanima W. Myeloproliferative neoplasms: trends in incidence, prevalence and survival in Norway. Eur J Haematol. 2017 Jan;98(1):85-93. doi: 10.1111/ejh.12788. Epub 2016 Sep 4. PMID 27500783
- [Background] Arber DA, Orazi A, Hasserjian R, et al. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016;127(20):2391-2405. Blood. 2016 Jul 21;128(3):462-463. doi: 10.1182/blood-2016-06-721662. No abstract available. PMID 31659364
- [Background] Linardi Cda C, Pracchia LF, Buccheri V. Diagnosis and treatment of polycythemia vera: Brazilian experience from a single institution. Sao Paulo Med J. 2008 Jan 2;126(1):52-7. doi: 10.1590/s1516-31802008000100010. PMID 18425288